CLINICAL TRIAL: NCT01792726
Title: An International Randomised Controlled Trial to Compare Targeted Intra-operative Radiotherapy Boost With Conventional External Beam Radiotherapy Boost After Lumpectomy for Breast Cancer in Women With a High Risk of Local Recurrence.
Brief Title: A Comparison of Intra-operative Radiotherapy Boost With External Beam Radiotherapy Boost in Early Breast Cancer.
Acronym: TARGIT-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGIT Boost; NHS NIHR HTA (Other Grant/Funding Number: 10/104/07)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Early Breast Cancer
Keywords: breast cancer; radiotherapy; TARGIT; Intrabeam
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TARGIT (Experimental): The experimental policy is to give targeted intra-operative radiotherapy (TARGIT-Boost) in a single dose to substitute for the usual boost dose, in addition to whole breast external beam radiotherapy delivered according to local treatment guidelines.
  Interventions: Radiation: Boost to the tumour bed
- External beam radiotherapy boost (Active Comparator): The conventional policy is to receive radiation boost to the tumour bed delivered by external beam radiotherapy (EBRT) in addition to whole breast external beam radiotherapy delivered according to local treatment guidelines.
  Interventions: Radiation: Boost to the tumour bed

INTERVENTIONS:
Radiation: Boost to the tumour bed — Boost to the tumour bed, with whole breast EBRT delivered according to local policy.
  Other Names: Radiotherapy boost

SUMMARY:
TARGIT-Boost is an international randomised clinical trial designed to test the hypothesis that the tumour bed boost delivered as a single dose of targeted intraoperative radiotherapy (TARGIT-B) is superior to the conventional course of external beam radiotherapy boost (EBRT-Boost), especially in women with high risk of local recurrence. It is a pragmatic trial in which each participating centre can use the local predefined inclusion/exclusion criteria for entry into the trial. Only centres with access to the Intrabeam® (Carl Zeiss) are eligible to enter patients into the trial.

Eligible patients are those with a higher risk of local recurrence after breast conserving surgery.

After giving consent patients are randomised to either TARGIT Boost or EBRT Boost. All patients will receive whole breast EBRT. They may receive any other adjuvant treatments as deemed necessary. The protocol recommends that patients be followed at six monthly intervals for three years and then annually.

The primary endpoint is ipsilateral breast recurrence rate. Secondary endpoints are relapse-free survival, site of recurrence, overall survival (breast-cancer specific and non-breast cancer deaths) patient satisfaction and quality of life.

DETAILED DESCRIPTION:
DESIGN: A pragmatic multi-centre randomised clinical trial to test whether TARGeted Intraoperative radioTherapy as a tumour bed Boost (TARGIT-B) is superior in terms of local relapse within the treated breast compared with standard post-operative external beam radiotherapy boost in women undergoing breast conserving therapy who have a higher risk of local recurrence. Patients can be entered before the primary surgery or in a smaller proportion of cases, post-pathology. SETTING: Specialist breast units in UK, USA, Canada, Australia and Europe; 31 centres currently recruiting in the TARGIT-A trial and several are ready to join. TARGET POPULATION: Breast cancer patients suitable for breast conserving surgery, but with a high risk of local recurrence. Details of inclusion and exclusion are given in part 2. Briefly the patients should be either younger than 45 or if older, need to have certain pathological features that confer a high risk of local recurrence of breast cancer. HEALTH TECHNOLOGIES BEING ASSESSED. The TARGIT Technique: The Intrabeam® (Carl Zeiss, FDA approved and CE marked) is a miniature electron beam-driven source which provides a point source of low energy X-rays (50kV maximum) at the tip of a 3.2mm diameter tube. The radiation source is inserted into the tumour bed immediately after excision of the tumour and switched on for 20-35 minutes to provide intra-operative radiotherapy accurately targeted to the tissues that are at highest risk of local recurrence. The physics, dosimetry and early clinical applications of this soft x-ray device have been well studied. For use in the breast, the technique was first developed and piloted at University College London. The radiation source is surrounded by a spherical applicator, specially designed (and available in various sizes) to produce a uniform field of radiation at its surface, enabling delivery of an accurately calculated dose to a prescribed depth. It is inserted in the tumour bed and apposed to it with surgical sutures and/or other means. As the x-rays rapidly attenuate the dose to more distant tissues is reduced; this also allows it to be used in standard operating theatres. 20 Gy is delivered to the tumour bed surface in 20-35 minutes, after which the radiation is switched off, the applicator removed, and the wound closed in the normal way. This simple technique has potentially several advantages over convential external beam radiotherapy, interstitial implantation of radioactive wires or conformal external beam radiotherapy. The first pilot of twenty-five cases was at performed at UCL using TARGIT technique as a replacement for the boost dose of radiotherapy; full dose external beam treatment was subsequently given. The phase II study of 300 patients was published and recently updated with long term data along with favourable toxicity and cosmetic outcome results of individual cohorts. A mathematical model of TARGIT developed recently (funded by Cancer Research UK) suggests that it could be superior to conventional radiotherapy. Translational research has found that TARGIT impairs the surgical-trauma-stimulated proliferation and invasiveness of breast cancer cells. This effect of radiotherapy may act synergistically with its tumouricidal effect yielding a superior result. MEASUREMENT OF COST AND OUTCOME: Patient assessments will be clinical examination (6 monthly x 3 years then yearly x 10 years) and mammography (yearly). with ulstrasound (if needed) . Primary outcome: histologically/cytologically proven local recurrence. Secondary: site of relapse in the breast, overall survival, local toxicity (RTOG and LENT SOMA criteria), cosmesis, quality of life, patient satisfaction and health economics. The cost and cost-effectiveness of TARGIT versus EBRT, both as boost, will be calculated from a NHS and personal social services (PSS) perspective. Costs directly incurred by patients will also be assesed, since EBRT as a boost is likely to impose additional time and travel expense to patients and families.

ELIGIBILITY:
Inclusion Criteria:

At least one of these criteria must be satisfied:

1. Less than 46 years of age
2. More than 45 years of age, but with one of the following poor prognostic factors:

   1. lymphovascular invasion
   2. gross nodal involvement (not micrometastasis)
   3. more than one tumour in the breast but still suitable for breast conserving surgery through a single specimen
3. More than 45 years of age, but with at least two of the following poor prognostic factors

   1. ER and/or PgR negative
   2. Grade 3 histology
   3. Positive margins at first excision
4. Those patients with large tumours which have responded to neo-adjuvant chemo- or hormone therapy in an attempt to shrink the tumour and are suitable for breast conserving surgery as a result.
5. Lobular carcinoma or Extensive Intraductal Component (EIC)
6. A list (one to many) of high risk factors are present (as predefined in the policy document) that give a high risk of local recurrence.
7. Patients with either HER2 positive or HER2 negative can be included.

Exclusion Criteria:

1. Bilateral breast cancer at the time of diagnosis.
2. Patients with any severe concomitant disease that may limit their life expectancy
3. Previous history of malignant disease does not preclude entry if the expectation of relapse-free survival at 10 years is 90% or greater (e.g., non-melanoma skin cancer, CIN, etc).
4. No more than 30 days can have elapsed between last breast cancer surgery (not axillary) and randomisation for patients in the post-pathology stratification unless part of a specific clinical trial that addresses the question of timing or tumour bed can be reliably identified, e.g., by ultrasound.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1796 (Estimated)
Dates: Start 2013-06; Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Local tumour control (defined as no recurrent tumour in the ipsilateral breast). | Five year median follow-up
  To evaluate whether a tumour bed boost in the form of a single fraction of radiotherapy given intra-operatively and targeted to the tissues at the highest risk of local recurrence is superior (in terms of local tumour control) to standard post-operative external beam radiotherapy boost, after breast conserving surgery in women undergoing breast conserving therapy who have a higher risk of local recurrence.

SECONDARY OUTCOMES:
Site of relapse within the treated breast | 5 years median follow-up
  Site of relapse within the breast will be recorded in order to assess whether the recurrence is at the site of the initial tumour or at a new site and whether it has occurred within the treated field (TARGIT or EBRT boost).
Relapse-free survival | Five year median follow-up
  Relapse-free survival will be recorded as the time interval between randomisation and the date of confirmation of recurrence. The actual date to be used is the clinic day on which the investigations that led to a confirmed diagnosis of the recurrence were requested. Relapse-free survival will include any recurrence of breast cancer or death without a prior report of relapse.
Overall survival | Five year median follow-up.
  Overall survival will be the time interval between randomisation and death.
Adverse events related to the primary treatment of the breast cancer. | Five year median follow-up.
  Local toxicity and morbidity will be recorded as adverse events related to the primary treatment of the breast cancer. Quality of life will be assessed though validated patient-completed questionnaires.
Quality of life assessed by patient completed validated questionnaires. | Five year median follow-up
  The primary patient reported outcome endpoint for quality of life will be the FACT-B+4 trial outcome index (TOI) score. The TOI score (0-180) is a sum of the scores of the 27 items included in the physical well-being, functional well-being and breast cancer subscales of the FACT-B+4. A change of at least 5 points in TOI is considered to be clinically relevant or a minimally important difference (Eton et al. 2004). Secondary endpoints will be: 1) the five item arm functioning subscale score (0-20) 2) The 40 item FACT B+4 score (0-160), which reflects global quality of life including social and emotional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant S Vaidya, MBBS FRCS, Principal Investigator — University College, London
Locations (34):
- United States (8):
  - Helen Rey Breast Cancer Research Foundation, Los Angeles, California
  - Memorial Health University Medical Center, Savannah, Georgia
  - Beaumont Health - Royal Oak, Detroit, Michigan
  - Lakeland Regional Health System, Saint Joseph, Michigan
  - Ashikari Breast Center, Dobbs Ferry, New York
  - Cleveland Clinic, Cleveland, Ohio
  - West Virginia University, Morgantown, West Virginia
  - Aurora Breast Center, Green Bay, Wisconsin
- Beijing Cancer Hospital, Beijing, China
- France (7):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital Nord, Marseille
  - Institut de Cancerologie de l'Ouest site René Gauducheau, Nantes
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Italy (2):
  - Centro Di Riferimento Oncologico Di Aviano, Aviano
  - Istituto Oncologico Veneto, Padua
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- University of Dammam, Dammam, Saudi Arabia
- Netcare Milpark Hospital, Johannesburg, South Africa
- Gangnam Severance Hospital, Seoul, South Korea
- Spain (2):
  - Institut Català d'Oncologia, Barcelona
  - Hospital Universitario Dr Negrín, Las Palmas de Gran Canaria
- Brust-Zentrum Onkologie, Zurich, Switzerland
- Queen Sirikit Cantre for Breast Cancer, Bangkok, Thailand
- United Kingdom (8):
  - Princess Alexandra Hospital NHS Trust, Harlow
  - Whittington Hospital, London
  - Royal Free London NHS Trust, London
  - Guy's Hospital, London
  - Hospital of St John and St Elizabeth, London
  - Princess Grace Hospital, London
  - The Great Western Hospital, Swindon
  - Hampshire Hospitals NHS Foundation Trust, Winchester